CLINICAL TRIAL: NCT06583447
Title: Time Restricted Eating in Childhood Obesity: an Open-Label, Blinded-Endpoint, Parallel-Controlled, Randomized Clinical Trial
Brief Title: Time Restricted Eating in Childhood Obesity (TRECO)
Acronym: TRECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoyan Shi (Other)
Collaborators: Soochow University (Other)
Responsible Party: Sponsor-Investigator, Xiaoyan Shi, Associate Chief Physician, Children's Hospital of Soochow University
Organization: Children's Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRECO-suzhou; ChiCTR2400088243 (Other: ChiCTR)
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Calory-restricted diet; time-restricted eating
MeSH Terms: conditions — Pediatric Obesity; Intermittent Fasting | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRD group (Active Comparator): Based on the standardized lifestyle intervention, the study subjects in the control group will be treated with CRD. Total daily energy intake will be restricted to 80% of the energy requirement for each age group in the Dietary Reference Intakes of Nutrients for Chinese Residents DRIs 2013. A daily food diary will be kept at least one weekday and one weekend per week.
  Interventions: Behavioral: Calorie-restricted diet (CRD)
- TRE group (Experimental): Based on the standardized lifestyle intervention, TRE is administered to the study subjects in the intervention group. The eating window is limited to 12 hours per day, with the last meal no later than 7:00 p.m., and the study subjects are free to choose their eating window. Energy intake is not restricted during the eating period, and calorie-free, sugar-free beverages (water, tea, coffee) are allowed during the fasting period. A daily food diary will be kept for at least one weekday and one weekend per week.
  Interventions: Behavioral: Time-restricted eating (TRE)

INTERVENTIONS:
Behavioral: Calorie-restricted diet (CRD) — Standardized lifestyle interventions for all obese children and their parents will be constructed by endocrinologists and dietitians to increase physical activity and healthy eating habits. Physical activity interventions include decreasing time spent in sedentary activities, increasing the amount of physical activity, and recommending at least 60 minutes of moderate-intensity exercise per day. Individualized dietary counseling is provided to address the comorbidities in obese children.
  Based on the standardized lifestyle intervention, the study subjects in the control group will be treated with CRD. Total daily energy intake will be restricted to 80% of the energy requirement for each age group in the Dietary Reference Intakes of Nutrients for Chinese Residents DRIs 2013. A daily food diary will be kept for at least one weekday and one weekend per week.
  Arms: CRD group
Behavioral: Time-restricted eating (TRE) — Based on the standardized lifestyle intervention mentioned by the calorie-restricted diet (CRD) intervention, TRE is administered to the study subjects in the intervention group. The eating window is limited to 12 hours per day, with the last meal no later than 7:00 p.m., and the study subjects are free to choose their eating window. Energy intake is not restricted during the eating period, and calorie-free, sugar-free beverages (water, tea, coffee) are allowed during the fasting period. A daily food diary will be kept for at least one weekday and one weekend per week.
  Arms: TRE group

SUMMARY:
The goal of this clinical trial is to learn if time-restricted eating (TRE), an alternative method of reducing energy intake which has gained popularity in recent years, works to treat obesity in children. It will also learn about the safety and long-term adherence of 12-hour TRE, in comparison to calory restricted diet (CRD) . The main questions it aims to answer are:

1. Is the weight-losing effect of 12-hour TRE better than CRD?
2. Is 12-hour TRE easier to adhere to than CRD?

Researchers will compare 12-hour TRE to CRD (the primary treatment for obesity) to see if 12-hour TRE works to treat childhood obesity.

Participants will:

1. Follow the 12-hour TRE or CRD diet every day for 48 weeks;
2. Visit the clinic once every 4 weeks before 12 weeks and thereafter every 12 weeks for checkups and tests;
3. Keep a diary of their diet, physical activity, and symptoms

DETAILED DESCRIPTION:
Childhood obesity is a major metabolic disorder affecting approximately 20% of children and adolescents. Calory-restricted diet (CRD) is the primary treatment for obesity, but adherence to CRD typically declines over time and many individuals who lose weight with this strategy regain it. Accumulating evidence suggests that time-restricted eating (TRE), an alternative method of reducing energy intake that has gained popularity in recent years, has a significant weight-losing effect on adult obesity. However, its weight-losing effect on childhood obesity is still lacking trial evidence.

The overall objective of this study is to test the effectiveness of 12-hour TRE on weight loss for childhood obesity in comparison with CRD. The secondary objective is to compare the long-term adherence and weight-losing effect between the two dietary interventions.

The TRECO study is an open-label, blinded endpoint, parallel design, randomized controlled trial planned to enroll 128 patients with childhood obesity (8-17 years old, BMI-Z value >2), randomized by sex and age (12 years old) into zonal groups, and on the basis of the conventional non-pharmacological interventions, TRE was given to the intervention group, and CRD was given to the control group, and the short-term effect of TRE was observed after 12 weeks of intervention The short-term effect of TRE was observed after 12 weeks of intervention, i.e., to compare the difference in the magnitude of BMI-Z reduction between the two groups. The intervention was extended to 48 weeks to observe the long-term effect of TRE by comparing the difference in the reduction of BMI-Z between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age: 8-17 years.
* Childhood obesity: BMI-z score > 2.
* Agree to participate in this study and signed an informed consent form.

Exclusion Criteria:

* Individuals who have been actively fasting for more than 12 hours/day.
* Diabetic patients on hypoglycemic medications.
* Individuals undergoing weight loss interventions or previous bariatric surgery.
* Individuals with psychiatric, intellectual developmental disorders, or aphasia.
* Individuals on appetite or weight-suppressing medications within the last three months (e.g., antipsychotics, hypnotics, weight-loss drugs, insulin).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in BMI-Z score | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Weight and height are monitored at all-time points with an electronic scale and stadiometer and combined to calculate BMI-Z score based on the WHO growth charts. Participants will wear minimal clothing during the height and weight measurements.

SECONDARY OUTCOMES:
Weight attainment rate | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Weight and height are monitored at all-time points with an electronic scale and stadiometer and combined to calculate BMI-Z score based on the WHO growth charts. Participants will wear minimal clothing during the height and weight measurements. Weight attainment is defined as a BMI-Z score <2.
Change in body composition | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Body composition is assessed by bioimpedance with a Tanita MC-780 BC instrument, available at the Hospital's Endocrinology department. We are monitoring the absolute amount and percentage of both total body fat and lean mass as well as abdominal fat mass at all time points.
Quality of life | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Quality of life scale for children and adolescents (QLSCA), a multi-dimensional self-evaluation scale for learning and life, covering physical, psychological, social function and living environment, is suitable for primary and middle school students aged 7 to 18.
Sleep quality | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Sleep quality was assessed by a total score of the Pittsburgh Sleep Quality Index (PSQI).
Eating behavior | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Children eating behavior questionnaire (Children's Eating Behavior Questionnaire, CEBQ) using 35 items, 8 subscale to assess children's eating behavior habits. CEBQ measures food "close" (food response, food enjoyment, emotional overeating, drink desire) and food "avoidance" (satiety reaction, eating slowly, picky, and emotional deficiency) eating behavior.
Adherence | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Leveraging dietary diary, the compliance will be assessed by days when study subjects completed the dietary intervention program.
Energy intake | Every week from enrollment to the end of treatment at 48 weeks
  24 hour meal review through the whole study
Change in hemoglobin A1c | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Blood biochemical analyzer was used to detect hemoglobin A1c as the indicator of glucose metabolism.
Change in low density lipoprotein cholesterol | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Blood biochemical analyzer was used to detect low density lipoprotein cholesterol to assess lipids metabolism.
Change in systolic blood pressure | From enrollment to the end of treatment at 12 (stage 1) and 48 (stage 2) weeks respectively
  Sitting blood pressure was measured three times at resting state, with the mean as blood pressure. Systolic blood pressure was used to assess the blood pressure control..

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Children's Hopital of Soochow University, Suzhou, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
The protocol of this study will be published in open peer-reviewed journals very soon.

REFERENCES:
- [Background] Varady KA, Cienfuegos S, Ezpeleta M, Gabel K. Clinical application of intermittent fasting for weight loss: progress and future directions. Nat Rev Endocrinol. 2022 May;18(5):309-321. doi: 10.1038/s41574-022-00638-x. Epub 2022 Feb 22. PMID 35194176
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Juonala M, Magnussen CG, Berenson GS, Venn A, Burns TL, Sabin MA, Srinivasan SR, Daniels SR, Davis PH, Chen W, Sun C, Cheung M, Viikari JS, Dwyer T, Raitakari OT. Childhood adiposity, adult adiposity, and cardiovascular risk factors. N Engl J Med. 2011 Nov 17;365(20):1876-85. doi: 10.1056/NEJMoa1010112. PMID 22087679
- [Background] Bjerregaard LG, Jensen BW, Angquist L, Osler M, Sorensen TIA, Baker JL. Change in Overweight from Childhood to Early Adulthood and Risk of Type 2 Diabetes. N Engl J Med. 2018 Apr 5;378(14):1302-1312. doi: 10.1056/NEJMoa1713231. PMID 29617589